CLINICAL TRIAL: NCT05145244
Title: Copenhagen Master Observational Trial (C-MOT): A Prospective Investigator-initiated Observational Study to Study Biomarkers in Relation to Clinical Outcome in Patients With Non-Small Cell Lung Cancer or Breast Cancer
Brief Title: Copenhagen Master Observational Trial
Acronym: C-MOT
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulrik Lassen, Head of department, Rigshospitalet, Denmark
Other Study IDs: C-MOT
Record Dates: First submitted 2021-09-27; First posted 2021-12-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer; Breast Cancer
Keywords: Real world data; Observational trial; WGS, whole genome sequencing; Patient Reported Outcomes, PRO
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Diagnostic specimens will be used as baseline, and new biopsies will be performed at progression if feasible. A fresh tumor sample from metastatic sites will be obtained under local anaesthesia. If adequate tissue is available, samples are stored in RNAlater (Life Technologies) for RNA expression analyses and DNA gene mutation analyses and one sample is being formalin-fixed, paraffin-embedded (FFPE) for histopathologic analyses. Otherwise, formalin-fixed, paraffin-embedded (FFPE) will be used for WGS. A blood sample (7 mL EDTA) is collected for germline mutation analysis.
  Liquid biopsies will be performed at baseline and at every treatment cycle. Peripheral blood is collected in BCT tubes (Streck Laboratories, Omaha, NE, USA). Circulating DNA (cfDNA) will be extracted from 2-4 ml plasma using the QIAsymphony Circulating DNA Kit (Qiagen, Hilden, Germany).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with newly diagnosed non-small cell lung cancer: Approximately 1800 patients who are initiating
  * Standard of care, including targeted therapy based on PD-L1 status, EGFR, ALK or ROS1 (routine biomarkers)
  * Active clinical trials in the clinics after informed consent
  Interventions: Other: NO intervention
- Patients with metastatic breast cancer: Approximately 600 patients who are initiating
  * Standard of care, including targeted therapy based on HER2 status and ER status (routine biomarkers)
  * Active clinical trials in the clinics after informed consent
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — No intervention

SUMMARY:
The primary objectives of this prospective non-interventional study (NIS) are to assess and describe outcomes in relation to biomarkers, including whole-genome sequencing (WGS) in patients with non- small cell lung cancer (NSCLC) or breast cancer receiving treatment offered in the clinic (standard of care or included in clinical trials).

DETAILED DESCRIPTION:
To date, there have been few studies evaluating the day- to-day effects of non-small cell lung cancer (NSCLC), and advanced (ABC) or metastatic breast cancer (mBC) and its treatment on patients in a real-world setting. There is a gap between the data from the narrowly focused low-quantity, high-quality interventional studies and less granular data collection, high-quantity real world data (RWD). Therefore, prospective, observational trials including all patients independent of biomarkers and collecting comprehensive data on each are needed.

Research question and objectives:

* To describe treatment outcomes based on RWD by a complete set of clinical, socio-psychological, medico-economics data and biospecimens, including whole genome sequencing (WGS) of all patients with breast cancer and NSCLC.
* To record the treatment-related adverse events and late effects experienced by patients based on PRO tools.
* To perform refined biomarker analyses, including (but not limited to) whole genome sequencing, on tumor biopsies at baseline and at progression, in order to identify potential treatment targets.

Study design: Prospective, non-interventional, multicenter study of patients initiating treatment for NSCLC or breast cancer in Copenhagen (Denmark).

Population: Eligible patients will have breast cancer or NSCLC and acceptable performance status and organ function.

Data sources: Study data will be collected via a baseline site questionnaire; Patient Reported Outcomes (PRO) questions via mobile application at cycle-based intervals; and patient medical information from medical records into an eCRF at baseline and at every visit until the end of the follow-up period. Baseline WGS will be performed on diagnostic/surgical specimens after informed consent according to the Danish law of the National Genome Center. There are no specific protocol-mandated tests, procedures, or clinic visits for this study, but repeat sequential biopsies for WGS are optional at progression. All data collection for this study will occur over a 30-months period (including all treatment lines for new patients included in the period).

Study size: Up to 2400 patients diagnosed with NSCLC or breast cancer will be enrolled. Breast cancer patients will be enrolled at Rigshospitalet, and NSCLC at Rigshospitalet and Herlev Hospital. Any patient who meets the eligibility criteria will be invited to participate in the study. Eligibility will be assessed prior to enrollment during a scheduled visit.

Data analysis: Analyses will generally be descriptive and explorative in nature and will be conducted using SPSS statistical software, and no sample size calculations can be performed. All variables will be summarized descriptively through tabular displays of mean, median, ranges, and standard deviations of continuous variables and frequency distributions of categorical variables. Exploratory analyses may be conducted to examine correlations and/or other research questions (e.g., time-to-first-neutropenia using Kaplan- Meier methods or mutational status and response). No formal hypothesis testing or comparisons between treatment groups are performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥ 18 years of age) with diagnosis of NSCLC or breast cancer amenable to medical or radiation therapy with curative or palliative intent
* Evidence of a personally signed and dated informed consent form document indicating that the patient has been informed of all pertinent aspects of the study
* Able to read and understand Danish
* Willing and able to complete collection of data including WGS

Exclusion Criteria:

* Patient with breast cancer initiating adjuvant systemic therapy
* In the judgment of the investigator, the patient's life expectancy is fewer than 3 months at the time of diagnosis of NSCLC or breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have non-small cell lung cancer or breast cancer and acceptable performance and organ function
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 years
  Time from baseline to progression (measured using RECIST v1.1)
Patient reported outcomes | 3 years
  Health related quality of life. Two istruments will be used: EQ-5D-5L and EORTC QLQ-C30. The EQ-5D-5L will be administered at baseline and after each chemo cycle. The EORTC QLQ-C30 will be administered at baseline and 3 months after baseline.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Time from baseline to death or censoring
Treatment response | 3 years
  Treatment response will be measured using RECIST v1.1
Adverse events | 3 years
  Adverse events will be measured using a selection of instruments from the NCI PRO-CTCAE Measurement System (Danish version 1.0).
  For patients with lung cancer, the selection includes question #8, 9, 15, 16, 19, 20, 24, 46, 48, 52, 53, 54, 56 as well as free text entry.
  For patients with breast cancer, the selection includes question #8, 15, 39, 46, 48, 52, 53, 54, 56 as well as free text entry.
Late effects | 3 years
  Late effects will be measured using a selection of instruments from the NCI PRO-CTCAE Measurement System (Danish version 1.0).
  For patients with lung cancer, the selection includes question #8, 9, 15, 16, 19, 20, 24, 46, 48, 52, 53, 54, 56 as well as free text entry.
  For patients with breast cancer, the selection includes question #8, 15, 39, 46, 48, 52, 53, 54, 56 as well as free text entry.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided